CLINICAL TRIAL: NCT00706420
Title: Islet Transplantation Alone (ITA) in Patients With Difficult to Control Type I Diabetes Mellitus Using a Glucocorticoid-free Immunosuppressive Regimen
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01083; RR-01-002
Record Dates: First submitted 2008-06-25; First posted 2008-06-27 (Estimated); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus; Islet Transplantation Alone; Glucocorticoid-free Immunosuppressive Regimen
MeSH Terms: conditions — Diabetes Mellitus | interventions — Islets of Langerhans Transplantation; Immunosuppression Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Islet cell transplantation alone
  Interventions: Procedure: Islet Transplantation + Immunosuppression; Biological: Islet cell transplantation

INTERVENTIONS:
Procedure: Islet Transplantation + Immunosuppression — Islet Transplantation + Immunosuppression (Sirolimus/Tacrolimus, daclizumab)
Biological: Islet cell transplantation — Islet cell transplantation will occur through the portal vein.

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of islet cell transplantation alone (ITA) in patients with difficult to control type I diabetes. Difficult to control type 1 diabetes is defined as wide swings in blood glucose that disrupt the patient's life and result in frequent episodes of low blood glucose despite the proper use of standard insulin therapy and frequent blood glucose monitoring.

DETAILED DESCRIPTION:
Type 1 diabetes is associated with the damage of a specific cell subtype of pancreatic islets (clusters of cells in the pancreas that produce insulin and other metabolic hormones), which makes patients depend on an outside source of insulin. Despite insulin treatment, type 1 diabetes mellitus causes a significant risk of long-term problems, including damage to the heart, blood vessels, nerves, eyes and kidneys. The results of recent research studies suggest that these complications are caused by poor glucose control.

Transplantation of islets offers the prospect of good glycemic (blood glucose) control without the major surgical risks associated with whole pancreas transplant and may result in not needing any insulin injections. In 2000, a group of investigators in Edmonton, Canada showed that islet transplantation using a combination of anti-rejection drugs to help prevent the rejection of transplanted islets was effective in eliminating insulin intake in 7 subjects who were followed up to 20 months. After 5 years, more than 60 patients have been transplanted at Edmonton and only 1 in 10 remained off of insulin.

This study is being performed to confirm the results of the Edmonton study to see if islet transplantation alone (ITA) is a safe and effective way of treating subjects with type 1 diabetes. This study uses a few additional medications and vitamin supplements that were not included in the original Edmonton study. We hope this will improve the long-term outcome of islet transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Difficult to control Type 1 diabetes mellitus (defined above). Documentation of negative basal and stimulated C-peptide (a basal level of < 0.2 ng/ml before IV administration of 1 mg of glucagon, and a glucagon stimulated C-peptide < 0.8 ng/ml) and diagnosis of diabetes for at least 5 years. When possible, patients will be evaluated with continuous glucose monitoring (GlucoseSensor ®) to determine the frequency and extent of hypo- and hyperglycemic episodes.
* No evidence of chronic renal failure or significant proteinuria (serum creatinine < 1.6 mg/dl, creatinine clearance >80 ml/min, and albumin excretion </= 300 mg/24 hr).
* No evidence of liver disease (liver enzymes < twice the upper limit of normal for each of ALT and AST, bilirubin < 2 mg/dl, albumin > 3.5 g/dl, and PT and PTT </= 1.1 x the upper limit of normal).
* Frequent episodes of symptomatic hypoglycemia (i.e. loss of consciousness, headaches, anxiety, irritability, trembling, sweating) more than once per week, documented hypoglycemic unawareness (i.e. no adrenergic and/or neurogenic symptoms with blood glucose < 54 mg/dl) two or more times in the past two months, or hypoglycemic episodes that required the assistance of another person more than once per month or hospitalization more than once over the past 20 months.
* Ability to comply with post-transplant regimen, including immunosuppression, insulin pump therapy and metabolic testing. Patients will be required to perform self-monitoring of blood glucose a minimum of four times daily, and provide complete records of blood glucose levels and insulin doses.
* Ability to give informed consent.
* Age greater than or equal to 18 years or less than or equal to 65 years.

Exclusion Criteria:

* Significant liver disease (including elevation of liver enzymes > twice the upper limit of normal for each of ALT and AST, bilirubin > 2 mg/dl, albumin < 3.5 g/dl, liver masses, portal vein thrombosis, evidence of portal hypertension, or significant, untreated gallbladder disease (i.e. gallstones).
* Significant cardiovascular disease, including non-correctable coronary artery disease with ejection fraction < 50% and/or recent myocardial infarction (within last 12 months); extensive peripheral vascular disease not correctable by surgery or untreated proliferative retinopathy.
* Recent unresolved acute infection, or chronic infection, including tuberculosis, HIV, HBV, HCV, CMV or positive skin test for TB.
* Any history of malignancy, except squamous or basal skin cancer or in situ cancer of the cervix.
* Recent history of non-compliance, or inability to demonstrate capacity to comply with strict blood glycemic control and insulin pump therapy.
* Psychiatric illness that is untreated, or likely to interfere significantly with transplantation despite treatment.
* Presence of preformed antibodies on panel reactive antibody screening > 20%.
* Body mass index (BMI) greater than 30.
* Age less than 18 years or greater than 65 years.
* Presence of a chronic disease that must be chronically treated with one or more of the following medications: glucocorticoids, diazoxide, bumetanide, haloperidol, chlorpromazine, desipramine, doxepin, imipramine, isoproterenol, levodopa, morphine, L-asparaginase, cyclophosphamide, isoniazid, heparin, nalidixic acid, or any other agents that may adversely influence glycemic control and which may confound the interpretation of Graft Success post-transplant.
* Pregnant women, women intending future pregnancy, women of reproductive potential who are unable or unwilling to follow effective contraceptive measures for the duration of immunosuppressive therapy, and women presently breast feeding are ineligible due to the unknown effects of these drugs on the fetus and nursing infant.
* Active alcohol or substance abuse, including cigarette smoking (must be abstinent for > 3 months).
* Hyperlipidemia (total cholesterol > 260 mg/dl, LDL > 130 mg/dl, and/or triglycerides > 300 mg/dl) despite appropriate treatment.
* Anemia (Hgb < 12 g/dl) or other hematologic disorders that require medical attention.
* Increased risk of bleeding (platelet count < 80,000; INR > 1.5), other chronic hemostasis disorders, or treatment with chronic anticoagulant therapy (i.e. heparin or warfarin).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2004-04-07 (Actual); Primary Completion 2026-10-12 (Estimated); Study Completion 2026-10-12 (Estimated)

PRIMARY OUTCOMES:
Percent of subjects who have achieved insulin independence post transplant. | 3, 6, 12, and 24 months

SECONDARY OUTCOMES:
Stimulated C-peptide response >0.6 ng/ml | 3, 6, 12, and 24 months
Insulin use </=0.2units/kg/day | 3, 6, 12, and 24 months
Reduction/elimination of hypoglycemic episodes | 3, 6, 12, and 24 months
HgAlc</= 6.5% | 3, 6, 12, and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Fouad Kandeel, MD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

REFERENCES:
- [Background] Shapiro AM, Lakey JR, Ryan EA, Korbutt GS, Toth E, Warnock GL, Kneteman NM, Rajotte RV. Islet transplantation in seven patients with type 1 diabetes mellitus using a glucocorticoid-free immunosuppressive regimen. N Engl J Med. 2000 Jul 27;343(4):230-8. doi: 10.1056/NEJM200007273430401. PMID 10911004
- [Background] Ryan EA, Paty BW, Senior PA, Bigam D, Alfadhli E, Kneteman NM, Lakey JR, Shapiro AM. Five-year follow-up after clinical islet transplantation. Diabetes. 2005 Jul;54(7):2060-9. doi: 10.2337/diabetes.54.7.2060. PMID 15983207